CLINICAL TRIAL: NCT00928447
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Single-Center Study of the Intradermal Injection of rHuPH20 or Placebo in Subjects With Nickel Allergic Contact Dermatitis
Brief Title: Study of the Intradermal Injection of rHuPH20 or Placebo in Participants With Nickel Allergic Contact Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HALO-114-201
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Dermatitis, Allergic Contact
Keywords: rHuPH20; Recombinant Human hyaluronidase
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rHuPH20 (Experimental): Participant's upper back will be divided into 2 equal spaces and will receive Regimen 1 and 2 in 4 spaces respectively. In Regimen 1, a single row of 4 patches, each with the nickel sulfate concentration (NSC) (1, 2.5, or 5%) determined at screening, will be applied to the upper space at Day 1. After 48 hours, the patches will be removed and the reactions will be graded on the ICDRG scale. An ID injection containing rHuPH20 (3,000 Units [U]) will be administered once daily (QD) for 5 days at the center of each area of reaction. In Regimen 2, a single row of 4 sites in the lower space will be injected intradermally with drug rHuPH20 (3,000 U) at Day 1. Ten minutes after the injections, patches with the NSC (1, 2.5, or 5%) determined at screening will be applied to the injection sites. After 48 hours, the patches will be removed and the reactions will be graded on the ICDRG scale. As during pretreatment, an ID injection containing rHuPH20 will be then administered QD for 5 days.
  Interventions: Drug: rHuPH20
- Placebo (Placebo Comparator): Participant's upper back will be divided into 2 equal spaces and will receive Regimen 1 and 2 in 4 spaces respectively. In Regimen 1, a single row of 4 patches, each with the NSC (1, 2.5, or 5%) determined at screening, will be applied to the upper space at Day 1. After 48 hours, the patches will be removed and the reactions will be graded on the ICDRG scale. An ID injection containing placebo will be administered QD for 5 days at the center of each area of reaction. In Regimen 2, a single row of 4 sites in the lower space will be injected intradermally with placebo at Day 1. Ten minutes after the injections, patches with the NSC (1, 2.5, or 5%) determined at screening will be applied to the injection sites. After 48 hours, the patches will be removed and the reactions will be graded on the ICDRG scale. As during pretreatment, an ID injection containing placebo will be then administered QD for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rHuPH20 — 0.25 milliliter (mL) Intradermal (ID) syringe push bolus injection of rHuPH20
  Arms: rHuPH20
Drug: Placebo — 0.25 mL ID syringe push bolus injection of placebo control
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect and safety of rHuPH20 or placebo for the prevention and treatment of skin allergic reaction to nickel. The study drug and placebo will be administered by intradermal injection.

DETAILED DESCRIPTION:
This study will involve 2 regimens which will run in parallel. Each participant's upper back will be divided into 2 equal spaces for Regimen 1 and 2. Each of the 4 treatment sites in each space will be independently randomized to placebo or rHuPH20 treatment in a 1:1 ratio. Thus, each participant will serve as their own control. Regimen 1 will evaluate the treatment of cutaneous reactions to nickel and Regimen 2 will evaluate the prevention as well as the treatment of cutaneous reactions to nickel. At screening, the nickel sulfate concentration (1%, 2.5%, or 5%) applied to the skin of the upper back with a patch, that will cause no more than a ++ reaction according to the scale of the International Contact Dermatitis Research Group (ICDRG) will be determined. This concentration will be used to elicit cutaneous reactions during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Females 18-60 years of age. Females of child-bearing potential must use a standard and effective means of birth control for the duration of the study.
* Known contact dermatitis to nickel with a confirmed positive patch-test result to nickel sulfate.
* Intact normal skin without potentially obscuring tattoos, acne, dermatitis, pigmentation or lesions on the posterior aspect of the torso (back) in the area intended for allergen testing and dose administration.
* Vital signs (blood pressure [BP], heart rate [HR], temperature, respiratory rate) within normal range or, if out of range, assessed by the Investigator as not clinically significant and it is mutually agreed by both Investigator and sponsor medical monitor that the participant need not be excluded from the study for this reason.
* A negative serum or urine pregnancy test (if female of child-bearing potential) within 14 days of initial study drug administration.
* Participant should be in good general health based on medical history and physical examination, without medical conditions that might prevent the completion of study drug injections and assessments required in this protocol.
* Decision-making capacity and willingness and ability to comply with the requirements for full completion of the study.
* Signed, written Institutional Review Board (IRB)/Ethics Committee (EC)-approved informed consent.

Exclusion Criteria:

* Nickel allergen patch test greater than a ++ reaction.
* Participants who were treated with chemotherapy agents or systemic corticosteroids within the past 3 months.
* Use of topical steroids, antihistamines, or immunosuppressants used near the site of allergen testing/injection within 14 days.
* Use of oral antihistamines within 14 days of study conduct.
* Extensive ongoing outbreaks of contact dermatitis anywhere on the body.
* Pregnant or women who are breast-feeding.
* Participants with a current disease state that can affect immune response (for example, flu, cancer, human immunodeficiency virus [HIV]).
* Known allergy to any hyaluronidase or the ingredients in the dose preparation.
* History of autoimmune disorder.
* Participants with any other medical condition that, in the opinion of the investigator, might significantly affect their ability to safely participate in the study or affect the conduct of this study. Examples might include asthma, diabetes, heart disease, epilepsy, cancer, etc.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06-23 (Actual); Primary Completion 2009-09-13 (Actual); Study Completion 2009-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ikeadi M Ndukwu, M.D., MPH, Principal Investigator — Saint Anthony Memorial Research Center
Locations (1):
- Symbio Phase I Unit, Saint Anthony Memorial Research Center, Michigan City, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a known history of nickel allergy were recruited. At screening, the nickel sulfate concentration (1%, 2.5%, or 5%), applied to the skin of the upper back with a patch, that caused no more than a ++ reaction according to the scale of the International Contact Dermatitis Research Group (ICDRG) was determined. This concentration was used to elicit cutaneous reactions during the study period.
Pre-assignment Details: This study involved 2 regimens which ran in parallel. Each participant's upper back was divided into 2 equal spaces for Regimen 1 and 2. Each of the 4 treatment sites in each space was independently randomized to placebo or rHuPH20 treatment in a 1:1 ratio. Thus, each participant served as their own control.
Units Other Than Participants: Patch
Groups:
- Overall Study (rHuPH20 and Placebo): Participant's upper back was divided into two equal spaces and received Regimen 1 and 2 in 4 spaces respectively. In Regimen 1, a single row of 4 patches, each with the nickel sulfate concentration (1, 2.5, or 5%) determined at screening, was applied to the upper space at Day 1. After 48 hours (Day 3), the patches were removed and the reactions were graded on the ICDRG scale. A 0.25 milliliters (mL) intradermal injection containing rHuPH20 (3,000 units [U]) or placebo (excipient) was administered once daily for 5 days at the center of each area of reaction. In Regimen 2, a single row of 4 sites in the lower space was injected intradermally with 0.25 mL of study material drug rHuPH20 (3,000 U) or placebo (excipient), in a randomly assigned 2:2 ratio at Day 1. Exactly ten minutes after the injections, patches with the nickel sulfate concentration (1, 2.5, or 5%) determined at screening were applied to the injection sites. After 48 hours (Day 3), the patches were removed and the reactions graded on the ICDRG scale. As during pretreatment, a 0.25 mL intradermal injection containing rHuPH20 or placebo was then administered once daily for 5 days at the center of each area of reaction.
Period: Overall Study
Arm/Group | Overall Study (rHuPH20 and Placebo)
Started | 22; 176 Patch
Received at Least 1 Dose of rHuPH20 (One half of the participant's back received rHuPH20) | 21; 168 Patch
Received at Least 1 Dose of Placebo (One half of the participant's back received placebo) | 21; 168 Patch
Completed | 20; 160 Patch
Not Completed | 2; 16 Patch
Not completed — Withdrawal by Subject | 1
Not completed — Investigator's decision | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all enrolled participants.
Groups:
- Overall Study (rHuPH20 and Placebo): Participant's upper back was divided into two equal spaces and received Regimen 1 and 2 in 4 spaces respectively. In Regimen 1, a single row of 4 patches, each with the nickel sulfate concentration (1, 2.5, or 5%) determined at screening, was applied to the upper space at Day 1. After 48 hours (Day 3), the patches were removed and the reactions were graded on the ICDRG scale. A 0.25 mL intradermal injection containing rHuPH20 (3,000 U) or placebo (excipient) was administered once daily for 5 days at the center of each area of reaction. In Regimen 2, a single row of 4 sites in the lower space was injected intradermally with 0.25 mL of study material drug rHuPH20 (3,000 U) or placebo (excipient), in a randomly assigned 2:2 ratio at Day 1. Exactly ten minutes after the injections, patches with the nickel sulfate concentration (1, 2.5, or 5%) determined at screening were applied to the injection sites. After 48 hours (Day 3), the patches were removed and the reactions graded on the ICDRG scale. As during pretreatment, a 0.25 mL intradermal injection containing rHuPH20 or placebo was then administered once daily for 5 days at the center of each area of reaction.
Arm/Group | Overall Study (rHuPH20 and Placebo)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Reaction Scores Based Upon ICDRG Scoring Scale: Regimen 1
Description: Cutaneous reactions at the patch test sites were scored according to the ICDRG scoring scale as Grade 0 (-)= Negative reaction, Grade 1/2 (?)= Doubtful reaction; faint macular erythema only, Grade 1 (1+)= Weak (nonvesicular) positive reaction; erythema, infiltration, papules, vesicles, Grade 2 (2+): Strong (vesicular) positive reaction; erythema, infiltration, papules, vesicles, Grade 3 (3+): Extreme positive reaction; bullous reaction Grade NA (IR): Irritant reaction of different types. Participants with positive reaction scores (>= Grade 1) have been reported in this outcome measure.
Time Frame: Day 3 (48 hours post-dose after the patch removal for Regimen 1) up to Day 14
Population: The Evaluable population included all evaluable participants who had completed dosing (or prematurely discontinued the administration due to a toxicity) and had undergone sufficient assessments to allow an assessment of the tolerability of the administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study (rHuPH20 and Placebo)
Number analyzed (Participants) | 20
Participants
  rHuPH20 | 5
  Placebo | 9

2. Primary Outcome: Number of Participants With Positive Reaction Scores Based Upon ICDRG Scoring Scale: Regimen 2
Description: as for outcome 1
Time Frame: Day 3 (48 hours post-dose after the patch removal for Regimen 2) up to Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study (rHuPH20 and Placebo)
Number analyzed (Participants) | 20
Participants
  rHuPH20 | 3
  Placebo | 2

3. Secondary Outcome: Percentage of Participants With a >=1 Grade Change in ICDRG Score in at Least One Patch Region After Treatment With rHuPH20 or Placebo: Regimen 1
Description: Cutaneous reactions at the patch test sites were scored according to the ICDRG scoring scale as Grade 0 (-)= Negative reaction, Grade 1/2 (?)= Doubtful reaction; faint macular erythema only, Grade 1 (1+)= Weak (nonvesicular) positive reaction; erythema, infiltration, papules, vesicles, Grade 2 (2+): Strong (vesicular) positive reaction; erythema, infiltration, papules, vesicles, Grade 3 (3+): Extreme positive reaction; bullous reaction Grade NA (IR): Irritant reaction of different types.
Time Frame: Day 3 (48 hours post-dose after the patch removal for Regimen 1)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study (rHuPH20 and Placebo)
Number analyzed (Participants) | 20
percentage of participants
  rHuPH20 | 70
  Placebo | 75

4. Secondary Outcome: Percentage of Participants With a >=1 Grade Change in ICDRG Score in at Least One Patch Region After Treatment With rHuPH20 or Placebo: Regimen 2
Description: as for outcome 3
Time Frame: Day 3 (48 hours post-dose after the patch removal for Regimen 2)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study (rHuPH20 and Placebo)
Number analyzed (Participants) | 20
percentage of participants
  rHuPH20 | 95
  Placebo | 90

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as adverse events (AEs) with an onset during or following administration of the first dose of study drug. AEs were defined as any untoward medical occurrence in a participant administered study drug and that did not necessarily have a causal relationship with the study drug. SAEs were defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. Adverse Events were only monitored/assessed on the whole participant level irrespective of different treatment regimen. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Baseline up to Day 14
Population: The Safety population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study (rHuPH20 and Placebo)
Number analyzed (Participants) | 21
Participants
  TEAEs | 21
  SAEs | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 14
Description: The Safety population included all participants who received at least one dose of study drug. Adverse Events were only monitored/assessed on the whole participant level irrespective of different treatment regimen.
Arm/Group | Overall Study (rHuPH20 and Placebo)
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (rHuPH20 and Placebo) (N=21)
Injection site pain (General disorders) | 21
Injection site pruritus (General disorders) | 18
Injection site discomfort (General disorders) | 3
Injection site haematoma (General disorders) | 3
Injection site irritation (General disorders) | 3
Feeling hot (General disorders) | 1
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must submit a copy of the proposed publication to the Sponsor 30 days prior to date of submission for publication. They can request a delay of up to 90 days if it is determined there is any patentable subject matter or confidential Information. Sponsor can make changes to the communication to remove sponsor's confidential information from it prior to publication.

DOCUMENTS (2):
  • Study Protocol (2009-05-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT00928447/Prot_000.pdf
  • Statistical Analysis Plan (2009-10-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT00928447/SAP_001.pdf